CLINICAL TRIAL: NCT05430230
Title: N of 1 Pilot Study of Nonsteroidal Anti-inflammatory Drugs in People With Painful Knee Osteoarthritis
Brief Title: Study of Nonsteroidal Anti-inflammatory Drugs in People With Painful Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00215311
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis, responder
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Naproxen

STUDY DESIGN:
Intervention Model Description: Participants will be entered into the trial and have an initial blinded 2-week treatment period of either naproxen or placebo and then entered into an open washout period of 2 weeks. At the end of this washout, participants will then receive either naproxen or placebo for a further 2 week period followed again by a 2 week washout. This sequence will then be repeated (total of 4 treatment periods) such that all participants receive naproxen for 2 treatment periods and placebo for 2 treatment periods. The order of treatment will be randomized and the treatment allocation and IP will be blinded.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All medication will be prepared in capsules identical in appearance and weight.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cross-over Treatment: Initial treatment with naproxen (Experimental): There will be a 4 period cross-over: 2 weeks of treatment with IP, followed by 2 weeks of washout, and this repeated 3 more times. Treatment will be such that all participants will receive 2 treatment periods with naproxen and 2 treatment periods with placebo. The order of treatment will be randomized and the treatment allocation and IP will be blinded.
  Interventions: Drug: Naproxen 500 Mg; Drug: Placebo
- Cross-over Treatment: Initial treatment with placebo (Experimental): There will be a 4 period cross-over: 2 weeks of treatment with IP, followed by 2 weeks of washout, and this repeated 3 more times. Treatment will be such that all participants will receive 2 treatment periods with naproxen and 2 treatment periods with placebo. The order of treatment will be randomized and the treatment allocation and IP will be blinded.
  Interventions: Drug: Naproxen 500 Mg; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen 500 Mg — naproxen tablets
  Other Names: non steroidal anti inflammatory drugs (NSAID)
Drug: Placebo — lactose NF

SUMMARY:
This is a pilot study with a 4-period double-cross-over design evaluating a treatment with non-steroidal anti-inflammatory drugs (NSAIDs) in people with painful knee osteoarthritis.

DETAILED DESCRIPTION:
Once screened and found eligible, participants will be entered into an initial blinded 2-week treatment period of either naproxen or placebo and then entered into an open washout period of 2 weeks. At the end of this washout, participants will then receive either naproxen or placebo for a further 2 week period followed again by a 2 week washout. This sequence will then be repeated (total of 4 treatment periods) such that all participants receive naproxen for 2 treatment periods and placebo for 2 treatment periods. The order of treatment will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >40 years of age
2. Meet ACR criteria for knee OA
3. Able and willing to provide informed consent
4. Average weekly pain in the index knee based on daily pain assessments of ≥ 4/10 and <9/10 on an 11-point NRS scale
5. Willing to discontinue current medications taken for OA pain
6. For women of child-bearing potential, willing to utilize some form of birth control or abstinence during the course of the study
7. If taking cannabinoids, have to be on a stable dose and have this maintained for the duration of the study
8. If receiving physical therapy or any non-pharmacologic modality(ies) for OA, these need to continue and remain stable for the duration of the study
9. Ambulatory
10. Have a cellphone and/or access to a computer and be able to utilize the eDiary as directed
11. Use of medications for knee OA pain on at least 4 out of 7 days per week
12. eDiary entries on at least 4 out 7 days per week during the observation period
13. Sub-Group Criterion (≥12 participants): Variability of average daily pain in the index knee during the observation period of ≥ 2 points on the NRS scale on at least 4 occasions

Exclusion criteria:

1. History of intolerance or allergic reaction to NSAIDs
2. Previous history of GI bleed
3. Renal insufficiency resulting in serum creatinine > 1.5 mg/dL
4. History of myocardial infarction in last 6 months
5. Coexisting congestive heart failure or symptomatic atherosclerotic heart disease
6. Use of oral anticoagulants other than aspirin ≤ 325 mg for cardiac prophylaxis
7. Use of heparin or injectable anticoagulant
8. Uncontrolled hypertension
9. Any medical condition which in the judgement of the investigator would make it inappropriate for the participant to enroll in the study
10. Use of recreational drugs
11. Fibromyalgia
12. Inflammatory arthropathies of any sort
13. Chronic back pain in which pain level is greater than the OA pain
14. Participation in another clinical trial other than one for covid or an observational and non-interventional study
15. Use of walker or other aid for walking other than a single cane
16. Hip pain on the ipsilateral side equal to or greater than the knee pain in the index joint
17. Index knee cannot have had previous joint replacement surgery
18. Arthroscopy within the past 6 months
19. Injection of hyaluronate in the index knee in the past 6 months
20. Corticosteroid injection in the index knee in the past 3 months
21. Injection of any biologic agent in the index in the past 12 months
22. Nerve ablation for the treatment of pain in the index knee
23. Any acute or chronic pain condition which would interfere with the evaluation of knee pain.
24. Pregnant, nursing or planning to become pregnant during length of study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean of one week's daily pain ratings on Numeric Pain Scale (NRS) 0-10; higher worse | baseline to end of 14 day treatment period
  daily pain will be collected by a web application and averaged over a 7day period; higher scores imply more pain

OTHER OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) 0-100; higher better | baseline to end of 14 day treatment period
  KOOS questionnaire
Pain Detect Questionnaire (PDQ) 0-38; higher more neuropathic | baseline to end of 14 day treatment period
  PDQ
Positive and Negative Affect Schedule (PANAS) questionnaire 10-50; higher more positive or negative affect | baseline to end of 14 day treatment period
  positive and negative affect
Quantitative Sensory Testing (QST) 0-100; higher is greater pain | baseline to end of 14 day treatment period
  quantitative sensory testing parameters - temporal summation
Oswestry Disability Index (ODI) 0-50; higher is greater disability | baseline to end of 14 day treatment period
  Oswestry Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No